CLINICAL TRIAL: NCT03652454
Title: Efficiency Of Micro-osteoperforation During Alignment Stage
Brief Title: The Evaluation Of The Efficiency Of Micro-osteoperforation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Asli Baysal, Assoc. Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016TDRSABE0026
Record Dates: First submitted 2017-10-18; First posted 2018-08-29 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Crowding of Teeth
Keywords: regional acceleratory phenomenon; micro-osteoperforation; orthodontic alignment
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Outcomes Assessor
Masking Description: single outcome assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- micro-osteoperforation (Experimental): Propel device (ABD) Micro-osteoperforations were performed in the keratinized tissue. Micro-osteoperforations were 1.5 mm in diameter and 3-7 mm in depth.
  Interventions: Device: micro-osteoperforation; Other: conventional fixed appliance treatment
- conventional treatment (Other): conventional fixed appliance treatment
  Interventions: Other: conventional fixed appliance treatment

INTERVENTIONS:
Device: micro-osteoperforation — Propel device (ABD) using for regional acceleratory phenomenon
  Arms: micro-osteoperforation
Other: conventional fixed appliance treatment — conventional fixed appliance treatment

SUMMARY:
Prolonged orthodontic treatment increases the risc of caries, periodontal problems and root resorption. Many different techniques were developed to shorten the treatment time. The aim of this study was to evaluate the effectiveness of micro-osteoperforations (MOP) performed in the alignment stage.

Twenty eight patients with mandibular arch discrepancy will be included in this research. After the patients are informed about the study they will be requested to sign the consent form.. At the beginning of the treatment routine orthodontic records (photographs, dental models and radiographs) will be taken and the gingival pocket measurements will be made.

The twenty eight patients will be randomly divided in two groups. In the first group, 3 or 4 micro-osteoperforations will be made in the parts of the gingiva nearby the discrepancy by perforating the keratinized or non-keratinized mucosa and reaching the alveolar bone under local anesthesia. In the further appointments the traditional aligning procedures will be used and controls will be made every 7-9 days. In the other group 20 patients will be treated in the traditional way and controls will be made each month. Every patient will be requested to answer questions related to treatment comfort and other problems like pain within the first week after each activations. The records will be repeated after the leveling phase. Tooth movement rate will be calculated according to the measurements made on dental casts. Measurements related to cephalometrics and gingival thickness will be evaluated. The results of two groups will be compared in terms of tooth movement rate, gingival thickness, pain and patient comfort.

DETAILED DESCRIPTION:
Twenty eight patients who have crowding in mandibular arch will be included in the study.

At the beginning of the study, routine orthodontic records and gingival measurements will be taken.All the records will be repeated after alignment stage.

Clinical periodontal parameters including plaque index, gingival index, pocket depth and bleeding were measured with Williams periodontal scaler (Hu Friedy®, Chicago, IL, USA).

Gingival thickness will be recorded with a ultrasonic device (Pirop® Ultrasonic Biometer A- Scan, Echo-Son, Krancowa, Poland) Irregularity index will be calculated for each patient using dental casts. After bracket placement; twenty eight patients will be randomly allocated to treatment and control groups (fourteen patients in each group) While micro-osteoperforations will be applied to treatment group, the control group will receive no additional treatment.

Each patient will be asked to fulfill a questionnaire to evaluate patient satisfaction and ease of operation.

The data was analyzed statistically and the level of statistical significance was determined as p ≤ .05.

ELIGIBILITY:
inclusion Criteria:

1. Existence of all permanent teeth (except molars 2 and 3)
2. Subjects aged 30 and below
3. Confusion of less than 8 mm according to model analysis of the upper and lower sieves
4. Gingival and periodontal indices of less than 1
5. Good oral hygiene

Exclusion Criteria:

1. Congenitally missing tooth
2. Severe skeletal malocclusion
3. Systemic disease affecting tooth movement
4. Active periodontal disease
5. Smoking
6. Radiographically detected bone loss
7. Gingival pocket depth greater than 4 mm
8. Previous surgical periodontal or orthodontic treatment

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Baysal, PhD, Study Director — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, İzmirli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faik Sahin M, Baysal A. The effect of micro-osteoperforation on the rate of tooth movement during the alignment stage in patients with mandibular crowding: a randomised controlled trial. Eur J Orthod. 2023 Sep 18;45(5):505-516. doi: 10.1093/ejo/cjad017. PMID 37167078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Micro-Osteoperforation, Regional Acceleration Phenomenon, Orthodontic Alignment
  Inclusion Criteria:
  * All permanent teeth have been worn (except 3rd molar)
  * More than 5 mm perforation compared to LII
  * Gingival and periodontal indices less than 1
  * Good hygiene
Groups:
- Micro-osteoperforation: Propel device (ABD)
  micro-osteoperforation: Propel device (ABD) using for regional acceleratory phenomenon. Propel® is a single-use device specially produced for micro-osteoperforation. The device contains a 1.5 mm thick perforation tip. It has a depth adjustment of 3, 5 and 7 mm and the LED depth indicator gives a warning when the desired depth is reached. The device was removed from its sterile packaging and, after setting the desired depth, was gently placed on the gum and turned clockwise with a slight pressure. When the desired skin was reached, it was removed by turning counterclockwise with the LED indicator on. Micro-osteoperforations were performed directly and atraummatically in the keratinized gum from two or three points, 3 mm between canine canine, 5 mm between canine molar, and 7 mm deep in the posterior region and 1.5 mm in diameter in the alveolar bone. The procedure was applied at the beginning of the study in the areas of crowding and not repeated.
- Conventional Treatment: conventional fixed appliance treatment
  conventional fixed appliance treatment: conventional fixed appliance treatment. Leveling with 0.014 inch nickel titanium (Ni-Ti, American Orthodontics, Sheboygan, WI, USA) arc wire was started in patients in each group using traditional fixed orthodontic bracket. All patients were invited to the controls once a month and each session was measured and a plaster model was created until the leveling phase was completed. Depending on the leveling, 0.014 inch, 0.016 inch, 0.016x0.022 inch and finally 0.019x0.025 inch Ni-Ti (American Orthodontics, Sheboygan, WI, USA) wires were used respectively. In both groups, arc wires were connected to the slots with prefabricated steel wire ligatures.
Period: Overall Study
Arm/Group | Micro-osteoperforation | Conventional Treatment
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The patients who have little irregularity index is more than 5 mm in the mandibular arches
Groups:
- Micro-osteoperforation: Propel device (ABD)
  micro-osteoperforation: Propel device (ABD) using for regional acceleratory phenomenon. Propel device (ABD)
  micro-osteoperforation: Propel device (ABD) using for regional acceleratory phenomenon. Propel® is a single-use device specially produced for micro-osteoperforation. The device contains a 1.5 mm thick perforation tip. It has a depth adjustment of 3, 5 and 7 mm and the LED depth indicator gives a warning when the desired depth is reached. The device was removed from its sterile packaging and, after setting the desired depth, was gently placed on the gum and turned clockwise with a slight pressure. When the desired skin was reached, it was removed by turning counterclockwise with the LED indicator on. Micro-osteoperforations were performed directly and atraummatically in the keratinized gum from two or three points, 3 mm between canine canine, 5 mm between canine molar, and 7 mm deep in the posterior region and 1.5 mm in diameter in the alveolar bone.
- Conventional Treatment: conventional fixed appliance treatment
  conventional fixed appliance treatment: conventional fixed appliance treatment conventional fixed appliance treatment
  conventional fixed appliance treatment: conventional fixed appliance treatment. Leveling with 0.014 inch nickel titanium (Ni-Ti, American Orthodontics, Sheboygan, WI, USA) arc wire was started in patients in each group using traditional fixed orthodontic bracket. All patients were invited to the controls once a month and each session was measured and a plaster model was created until the leveling phase was completed. Depending on the leveling, 0.014 inch, 0.016 inch, 0.016x0.022 inch and finally 0.019x0.025 inch Ni-Ti (American Orthodontics, Sheboygan, WI, USA) wires were used respectively. In both groups, arc wires were connected to the slots with prefabricated steel wire ligatures.
- Total: Total of all reporting groups
Arm/Group | Micro-osteoperforation | Conventional Treatment | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 12 | 23
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 14 | 14 | 28
little irregularity index [Mean (Standard Deviation); unit: millimetres] — Irregularity index is used to calculate the amount of crowding in the dental arches and measured in millimeters.
  There is no need to compare the measure with a standart or a norm (and neither according to sex or race or age).
  Generally crowding lower than 4 mm is classified as mild, crowding between 4-8 mm called moderate and crowding above 8 mm classified as severe.
  millimetres | 9.99 (2.63) | 8.87 (1.5) | 9.42 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Mandibular Teeth Alignment
Description: tooth movement rate (mm/month) was calculated. From the initiation of the treatment to the completion of alignment stage (approximately 6 months). All tooth movement rate measurements were performed in each month.
Time Frame: From the initiation of the treatment to the completion of alignment stage (approximately 6 months)
Population: * All permanent teeth have been erupted (except the 3rd molars)
  * Presence of more than 5 mm crowding in the lower arc according to Little irregularity index
  * Gingival and periodontal indices less than 1
  * Good oral hygiene
  * Patient and / or guardian volunteering to participate in the study
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Micro-osteoperforation: Propel device (ABD)
  micro-osteoperforation: Propel device (ABD) using for regional acceleratory phenomenon
Arm/Group | Micro-osteoperforation | Conventional Treatment
Number analyzed (Participants) | 14 | 14
millimeter (mm)
  first month | 4.27 (1.75) | 2.82 (0.87)
  second months | 2.08 (0.91) | 2.31 (1.29)
  third months | 1.94 (0.99) | 1.54 (0.65)
  fourth months | 0.84 (0.95) | 0.89 (0.49)
  fifth months | 0.34 (0.57) | 0.93 (0.7)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse effect were seen
Arm/Group | Micro-osteoperforation | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03652454/Prot_004.pdf
  • Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03652454/SAP_005.pdf